CLINICAL TRIAL: NCT01576536
Title: Genetic Variation in Platelet Aggregation
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 111760
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Platelet aggregation; cold pressor test; Genetics
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA and plasma/serum for subsequent biomarker analysis if required.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Normal healthy volunteers

SUMMARY:
The aim of the study is to test whether genetic variation in the alpha 2A adrenergic receptor affects diurnal variation in platelet aggregation.

DETAILED DESCRIPTION:
There is a marked diurnal fluctuation in the occurrence of acute myocardial infarction and sudden death, with peak incidences occurring in the early morning. Platelet aggregation has also been shown to increase in the early morning. The investigators will test the hypothesis that alpha 2a-adrenergic receptor (ADRA2A) genetic variation, specifically haplotype 4, affects platelet aggregation. The investigators will compare diurnal platelet aggregation in haplotype 4 subjects with subjects in the other haplotype families. In addition, the investigators will compare platelet aggregation after the cold pressor test in haplotype 4 with the other haplotype families. If there are no differences among haplotypes, then the haplotypes will be combined to analyze.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 45 years inclusive.
* Women of the above age will be studied between day 1 and day 14 of a normal menstrual cycle.
* Subjects must be willing to give informed consent for the study and able to adhere to the study diet and study procedures.
* Subjects and immediate extended family up till grandparents will be Caucasians or African Americans only.
* Subjects will be free of any clinically significant disease.
* Clinical laboratory test (CBC, blood chemistry) will be within acceptable limits.

Exclusion Criteria:

* Subjects who have taken any antiplatelet, anticoagulant or procoagulant medicines within the last three weeks preceding the study.
* Subjects who have taken medications (including over the counter medications) other than oral contraceptives in the past two weeks.
* Subjects who smoke or have smoked in the past 3 months.
* Subjects who are presently or were formerly a narcotic addict or alcoholic.
* Females with a positive pregnancy test.
* Females who are breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects will be recruited by advertisement and word-of-mouth.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MBChB, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- the Vanderbilt University General Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
all IDP that underlie results in a publication
Time Frame: 6 months after publication
Access Criteria: Access Criteria:
  IPD will be shared on request made to the PI. Criteria: Data is not to be shared. Data should only be used for biomedical research. Researchers requesting access will need appropriate IRB approval and sign a data use agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy normotensive, non-smokers Caucasians and African-Americans aged 18-45 years were recruited via flyers and word of mouth from 2012-2015. No medications except oral contraceptives within two weeks and no antiplatelet medications within three weeks of the study. Women were studied in the first 14 days of their menstrual cycle.
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 117
Completed | 117
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 37
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 117

OUTCOME MEASURES:

1. Primary Outcome: LogEC50 Platelet Aggregation
Description: EC50 represents the epinephrine concentration that produced 50% of maximal platelet aggregation (representing sensitivity to epinephrine) EC50 values were not normally distributed and were log-transformed for analyses.
Time Frame: at 6am and 930am
Population: outcome data could not be collected on all subjects, since unable to draw enough blood at a particular timepoint
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 108
nM
  LogEC50 at 6am | 2.65 (0.49)
  LogEC50 at 930am | 2.62 (0.44)

2. Secondary Outcome: Percentage, Adenosine Diphosphate (ADP) Induced Platelet Aggregation
Description: Blood samples were taken from participants and centrifuged. Adenosine Diphosphate (ADP) at a fixed concentration of 2.5 uM was added. Agonist-induced platelet aggregation was expressed as the percentage aggregation after 6 minutes of stimulation.
Time Frame: at 6am and 930am
Population: some outcome data could not be collected for all subjects, unable to draw enough blood for a particular timepoint
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 108
percentage of aggregation
  % aggregation at 6am | 72.8 (14.9)
  % aggregation at 930am | 75.8 (12.8)

3. Secondary Outcome: Percentage, Collagen Induced Platelet Aggregation
Description: Blood samples were taken from participants and centrifuged. Collagen at a fixed concentration of 2.5 ug/ml was added. Agonist-induced platelet aggregation was expressed as the percentage aggregation after 6 minutes of stimulation.
Time Frame: at 6am and 930am
Population: Some outcome date could not be collected for all subjects, unable to draw enough blood at a particular time point.
Measure: Mean (Standard Deviation); unit: percentage of platelet aggregation
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 108
percentage of platelet aggregation
  % platelet aggregation at 6am | 84.3 (7.9)
  % platelet aggregation at 930am | 83.5 (7.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time participant was admitted to the Clinical Research Center the evening before the study, to the end of the study, a 24 hour period.
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 1/117
Other Adverse Events (participants affected / at risk) | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=117)
acute right groin pain (General disorders) | 1 (1) — Study volunteer experienced acute right groin pain. He was taken to the Emergency Department treated with painkillers--had normal X-ray and MRI showing normal appearance of hip. Discharged from ED on analgesics--ED diagnosis "acute right groin pain".

LIMITATIONS AND CAVEATS:
Healthy young subjects studied, thus findings may not apply to different populations. Plasma catecholamines are an indirect measure of sympathetic activity--norepinephrine spillover would be more precise, but is technically demanding, not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes